CLINICAL TRIAL: NCT03454282
Title: Impact of Dietary Intervention on Tumor Immunity: the DigesT Trial.
Acronym: DIgesT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Collaborators: National Health Research Institutes, Taiwan (Other); Centro de Investigación en Nanomateriales y Nanotecnología (CINN) (Unknown); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Martin-Luther-Universität Halle-Wittenberg (Other); University of Milan (Other)
Responsible Party: Principal Investigator, Filippo de Braud, Professor, Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INT157/17; B42F17000260006 (Other Grant/Funding Number: Italian Minister of Health)
Record Dates: First submitted 2018-01-29; First posted 2018-03-05 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Breast Cancer; Melanoma, Malignant
Keywords: Breast; Cancer; Malignant; Melanoma; Fasting Mimicking Diet (FMD); Tumor; Immunity; Metabolic Effects; Immunological Effects
MeSH Terms: conditions — Breast Neoplasms; Melanoma; Neoplasms

STUDY DESIGN:
Intervention Model Description: Clinical trials with a single arm and three cohorts of patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FMD Arm (Experimental): The intervention consists in 5-day FMD (Fasting Mimicking Diet) to be followed for one cycle (Cohorts A and B) or for 4 consecutive every-four week cycles postoperatively.
  Interventions: Other: FMD

INTERVENTIONS:
Other: FMD — The Fasting Mimicking Diet (or FMD) consists in a 5-day plant-based, low-calorie (about 600 Kcal on day 1, followed by about 300 KCal/day on days 2 to 5), low-carbohydrate low-protein diet
  Other Names: Fasting Mimicking Diet

SUMMARY:
This trial aims to assess the immunological and metabolic changes induced by the Fasting Mimicking Diet (FMD) in the pre-operative and post-operative setting in breast cancer and melanoma patients. Three cohorts of patients will be enrolled: 1) Cohort A: patients with resectable breast cancer (cT1N0M0 stage or cT1cN1M0-cT2cN0M0 stages not requiring pre-operative systemic treatment at the judgment of the investigator) who are candidate to curative surgery; 2) Cohort B: patients with malignant melanoma patients candidate to dissection of the lymph node basin because of a positive sentinel lymph node (stage IIIA-IIIB-IIIC); 3) Cohort C: patients with resected malignant melanoma (including radicalization and, in case, lymph node dissection) who are not candidate to any adjuvant treatment, but only to clinical and radiological follow-up (stage IIB-IIC). Patients in cohorts A and B will undergo one 5-days FMD cycle about 13-15 days before surgical removal of primary tumor (breast) or lymph nodes (breast, melanoma). Patients in cohort C will undergo 4 consecutive FMD cycles every 28 days, starting one month after surgery.

DETAILED DESCRIPTION:
Preclinical evidences suggest that reducing the concentration of blood metabolites and growth factors reduces the in vivo growth of several tumor models, while protecting normal tissues from the cytotoxic effects of chemotherapeutical treatments. In recent years, a plant-based, calorie-restricted, low-carbohydrate, low-protein diet, also known as Fasting Mimicking Diet (FMD), has been proposed as a potential anticancer dietary intervention. The FMD is safe when administered cyclically (every 21-28 days) to healthy volunteers, and is capable of significantly reducing the concentration of plasma glucose, serum insulin and IGF-1, while increasing levels of plasma IGFBPs and ketone bodies. The FMD has been shown to inhibit the in vivo growth of several tumor models, including breast cancer and melanoma mice models. The anticancer effects of the FMD are likely mediated by two concomitant mechanisms: 1) one direct anticancer effect that is mediated by the inhibition of energy production and anabolic pathways, such as protein and fatty acid synthesis, in cancer cells; 2) one indirect effect that is mediated by the activation of antitumor immunity, with the result of enhanced tumor infiltration by cytotoxic CD8+ T-lymphocytes and reduced infiltration by immunosuppressive populations. According to the currently accepted model, the anticancer and immunomodulatory effects of the FMD mostly derive from the reduction of circulating glucose, insulin and IGF-1 levels, and a parallel increase of ketone body and IGF-1 binding protein concentration. However, recent observations in healthy volunteers and cancer patients, suggest that FMD-mediated changes in many other metabolites, such as specific amino acids or fatty acids, could contribute to the cell-autonomous or immune-mediated anticancer effects of the FMD. While the study of the effects of the FMD in combination with standard treatments (e.g. chemotherapy, molecular targeted therapy) in advanced cancers represents the final objective of the ongoing studies, fully uncovering the metabolic and immunological effects of the FMD alone is essential to design future combination studies. From this perspective, the pre- and post-operative clinical settings in cancer patients who are not candidate to other medical treatments represent an ideal context to assess the effects of the FMD without other confounding factors. This trial primarily aims to assess the immunological and metabolic changes induced by the FMD in the pre-operative and post-operative setting in breast cancer and melanoma patients. Three cohorts of patients will be enrolled: 1) Cohort A: patients with resectable breast cancer (cT1N0M0 stage or cT1cN1M0-cT2cN0M0 stages not requiring pre-operative systemic treatment at the judgment of the investigator) who are candidate to curative surgery; 2) Cohort B: patients with malignant melanoma patients candidate to dissection of the lymph node basin because of a positive sentinel lymph node (stage IIIA-IIIB-IIIC); 3) Cohort C: patients with resected malignant melanoma (including radicalization and, in case, lymph node dissection) who are not candidate to any adjuvant treatment, but only to clinical and radiological follow-up (stage IIB-IIC). Patients in cohorts A and B will undergo one 5-days FMD cycle about 13-15 days before surgical removal of primary tumor (breast) or lymph nodes (breast, melanoma). Patients in cohort C will undergo 4 consecutive FMD cycles every 28 days, starting one month after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 and ≤ 75 years.
2. Evidence of a personally signed and dated informed consent document (ICD) indicating that the patient has been informed of all pertinent aspects of the study before enrollment and FMD prescription.
3. Willingness and ability to comply with the FMD protocol, the scheduled visits, treatment plans, laboratory tests and other procedures.
4. Histologically confirmed diagnosis of invasive breast cancer candidate to curative surgery (Cohort A), or resected malignant melanoma requiring dissection of the regional lymph node basin for sentinel lymph node involvement (Cohort B), or malignant melanoma treated with curative surgery (including, in case, lymph node removal and lymph node dissection) (Cohort C). For breast cancer patients, any biological subgroup (including estrogen receptor-positive, HER2-positive, triple-negative breast cancer) will be admitted; HER2-positive tumors will be defined on the basis of an IHC score of 3, or a score of 2 with ISH evaluation indicative of gene amplification.
5. Availability of archival FFPE tissue blocks of primary breast cancer (Cohort A) or melanoma (Cohort B, Cohort C).
6. Presence of an Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
7. Presence of adequate bone marrow and organ function as defined by the following laboratory values:

   * ANC ≥ 1.5 x 109/l
   * platelets ≥ 100 x 109/l
   * hemoglobin ≥ 9.0 g/dl
   * calcium (corrected for serum albumin) within normal limits or ≤ grade 1 according to NCI-CTCAE version 4.03 if not clinically significant
   * potassium within the normal limits, or corrected with supplements
   * creatinine < 1.5 ULN
   * blood uric acid < 10 mg/dl
   * ALT and AST ≤ 2.5 x ULN
   * total bilirubin < ULN except for patients with Gilbert syndrome who may only be included in the total bilirubin is < 3.0 x ULN or direct bilirubin < 1.5 x ULN
   * Albumin > 3 g/dL
8. Fasting glucose ≤ 200 mg/dl.
9. Total Cholesterol ≤ 300 mg/dl.
10. Triglycerides ≤ 300 mg/dl.
11. Female patients of childbearing potential must agree to sexual abstinence or to use two highly effective method of contraception throughout the study and for at least 30 days after the end of the FMD. Abstinence is only acceptable if it is in line with the preferred and usual lifestyle of the patient. Examples of contraceptive methods with a failure rate of < 1% per year include tubal ligation, male sterilization, hormonal implants, established, proper use of combined oral or injected hormonal contraceptives, and certain intrauterine devices. Alternatively, two methods (e.g., two barrier methods such as a condom and a cervical cap) may be combined to achieve a failure rate of < 1% per year. Barrier methods must always be supplemented with the use of a spermicide. A patient is of childbearing potential if, in the opinion of the Investigator, she is biologically capable of having children and is sexually active.

Female patients are not of childbearing potential if they meet at least one of the following criteria:

* Have undergone a documented hysterectomy and/or bilateral oophorectomy
* Have medically confirmed ovarian failure
* Achieved post-menopausal status, defined as: (≥ 12 months of non-therapy-induced amenorrhea) or surgically sterile (absence of ovaries) and have a serum FSH level within the laboratory's reference range for postmenopausal females.

Exclusion Criteria:

1. Prior systemic treatment for breast cancer or melanoma.
2. Diagnosis of a concurrent malignancy other than breast cancer or melanoma, or malignancy other than breast cancer or melanoma diagnosed within 5 years of treatment enrollment, with the exception of adequately treated, basal or squamous cell carcinoma, non-melanomatous skin cancer or curatively resected cervical cancer.
3. Body Mass Index (BMI) < 20 Kg/m2.
4. Anamnesis of alcohol abuse.
5. Unintentional weight loss ≥ 5% in the last three months, unless the patient has a BMI > 25 Kg/m2 at study enrollment. Intentional weight loss is permitted if < 10% in the last three months and patient BMI is > 22 kg/m2.
6. Severe heart, liver, pulmonary, kidney comorbidities.
7. Current status of pregnancy or lactation, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test (> 5 mIU/mL).
8. Active HBV or HCV infection.
9. Severe infections within 4 weeks prior to FMD initiation, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia.
10. Active autoimmune diseases that require systemic treatment (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs).
11. History of recent diagnosis of hypothyroidism for which replacement therapy (eg., thyroxine) and blood endocrine profile are not stabilized yet.
12. Established diagnosis of diabetes mellitus type I or diabetes mellitus type II that requires pharmacological treatment (including, but not limited to, insulin, insulin secretagogues and metformin).
13. Severe impairment of the gastrointestinal (GI) function or GI disease that may alter the digestion and absorption of nutrients during the re-feeding phase (e.g. active ulcerative diseases of the stomach or intestine, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection).
14. Known history of Human Immunodeficiency Virus (HIV) infection.
15. Clinically significant heart disease and/or recent cardiac events including:

    * history of angina pectoris, coronary artery bypass graft (CABG), symptomatic pericarditis, or myocardial infarction within 12 months prior to the start of study treatment;
    * history of documented congestive heart failure (NYHA III-IV);
    * documented cardiomyopathy.
16. History of cardiac arythmias, (e.g. ventricular tachycardia, chronic atrial fibrillation), complete left bundle branch block, high grade AV block (e.g. bifascicular block, Mobitz type II and third degree AV block), supraventricular, nodal arrhythmias, or conduction abnormality in the previous 12 months.
17. Uncontrolled hypertension defined by a Systolic Blood Pressure (SBP) ≥ 160 mmHg and/or Diastolic Blood Pressure (DBP) ≥ 100 mmHg, with or without anti-hypertensive medication.
18. Known reduction of left-ventricular ejection fraction (LVEF) to less than 50%, as assessed by multigated radionuclide scintigraphic scan (MUGA) or echocardiography.
19. Previous episodes of symptomatic hypotension causing unconsciousness.
20. Baseline fasting plasma glucose ≤ 65 mg/dl.
21. Ongoing therapy with systemic corticosteroids, or systemic corticosteroid therapy ≤ 2 weeks before study enrollment, or who have not recovered from side effects of such treatment. The following uses of corticosteroids are permitted: topical applications (e.g. for rash), inhaled sprays (e.g. for obstructive airways diseases), eye drops.
22. Any serious medical or psychiatric illness that in the assessment of the investigator renders the patient not suitable for participation in this clinical study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2020-05-30 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Absolute and relative changes in PBMCs | 3 years
  Absolute and relative changes in PBMCs by 10-color cytofluorimetry before and after the FMD.

SECONDARY OUTCOMES:
Phenotypic modifications in PBMCs | 3 years
  Phenotypic modifications in PBMCs, as detected by by 10-colors citofluorimetry and single-cell "mass cytometry" (CyTOF)
Functional modifications in PBMCs | 3 years
  Functional modifications in PBMCs, as detected by by 10-colors citofluorimetry and single-cell "mass cytometry" (CyTOF)
Functional modifications in tumor-infiltrating lymphocytes | 3 years
  Functional modifications in tumor-infiltrating lymphocytes, as detected by by 10-colors citofluorimetry and single-cell "mass cytometry" (CyTOF)
Phenotypic modifications in tumor-infiltrating lymphocytes | 3 years
  Phenotypic modifications in tumor-infiltrating lymphocytes, as detected by by 10-colors citofluorimetry and single-cell "mass cytometry" (CyTOF)
Functional modifications of immune cell population in LNs | 3 years
  Functional modifications of immune cell populations in LNs, as detected by single-cell "mass cytometry" (CyTOF).
mRNA profiling in tumor cells | 3 years
  Gene expression profiling (through mRNA quantification) in tumor cells (Cohort A).
mRNA profiling in immune cells | 3 years
  Gene expression profiling (through mRNA quantification) in PBMCs and immune cell populations inside lymph nodes (Cohort B).
miRNA profiling in tumor cells | 3 years
  miRNA profiling in tumor cells (Cohort A)
miRNA profiling in immune cells | 3 years
  miRNA profiling in PBMCs and immune cell populations inside lymph nodes (Cohort B).
Changes in the expression of metabolic genes in PBMCs | 3 years
  Changes in the expression of selected metabolic genes (including hexokinase 1, phosphofructokinase 1, pyruvate kinase 2) through mRNA quantification in PBMCs before and after the FMD.
FMD-induced changes in blood metabolic parameters | 3 years
  FMD-induced changes in blood (glucose, triglycerides, fatty acids, cholesterol, amino acids)
FMD-induced changes in urine metabolites | 3 years
  FMD-induced changes in urine metabolites (ketone bodies)
FMD-induced changes in serum growth factors. | 3 years
  FMD-induced changes in serum growth factors.
Qualitative changes in tumor-infiltrating immune cells | 3 years
  Qualitative changes in the type of tumor-infiltrating immune cell populations before and after the diet in breast cancer patients undergoing curative surgery (Cohort A).
Quantitative changes in tumor-infiltrating immune cells | 3 years
  Quantitative changes in the number of tumor-infiltrating lymphocytes, machrophages, MDSCs before and after the diet in breast cancer patients undergoing curative surgery (Cohort A).
Changes in tumor proliferation | 3 years
  Changes in tumor proliferation index (Ki67) IHC in breast cancer patients (Cohort A).
Changes in tumor cell apoptosis | 3 years
  Changes in tumor cell apoptosis (caspase 3 by IHC) in breast cancer patients (Cohort A).
Changes in tumor metabolic pathways | 3 years
  Changes in tumor levels of glycolytic enzymes by IHC (Glut1, HK1, PFK1/2, PK2) in breast cancer patients (Cohort A).
Changes in expression of hormone receptors and HER2 | 3 years
  Changes in expression of estrogen and/progesterone receptor and HER2 oncoprotein by IHC in breast cancer patients (Cohort A).
Qualitative changes in immune cell suspensions from lymph nodes | 3 years
  Changes in the type of immune cells (CD8+ T-lymhocytes, CD 4+ lymphocytes, Treg) found in lymph node suspensions of melanoma patients undergoing one FMD cycle before lymph node dissection (Cohort B).
Quantitative changes in immune cell suspensions from lymph nodes | 3 years
  Quantitative changes in the absolute and relative amount of immune cell populations in lymph node suspensions of melanoma patients undergoing one FMD cycle before lymph node dissection (Cohort B).
Changes in DNA methylomic profiles in lymph node specimens | 3 years
  Changes in genome-wide DNA methylomic profiles with high-density arrays in lymph node specimens from patients undergoing the FMD before surgery (Cohorts A and B).
Changes in DNA methylomic profiles in tumor specimens | 3 years
  Changes in genome-wide DNA methylomic profiles with high-density arrays in tumor specimens from patients undergoing the FMD before surgery (Cohorts A and B).
Changes in gut microbiota composition. | 3 years
  Changes in type of gut bacteria populations, as detected through 16S ribosomal RNA sequencing
Short-term modification of blood nutritional parameters. | 3 years
  Short-term (before vs after each FMD cycle) modification of blood nutritional parameters (levels of plasma cholesterol, prealbumin, transferrin, total lymphocytes)
Long-term modification of blood nutritional parameters. | 3 years
  Long-term (along subsequent FMD cycles) modification of blood nutritional parameters (levels of plasma cholesterol, realbumin, transferrin, total lymphocytes)
Short-term and long-term modification of BMI | 3 years
  Short-term and long-term modification of BMI
FMD-induced changes in white blood cell populations | 3 years
  FMD-induced changes in neutrophils, macrophages, lymphocytes
FMD-induced changes in hemoglobin | 3 years
  FMD-induced changes in hemoglobin
Assessment of patient compliance to the FMD. | 3 years
  Assessment of patient compliance to the FMD, as measured by quantifying the number of major and minor deviations of patients' diet relative to the prescribed FMD scheme
Assessment of FMD tolerability. | 3 years
  Assessment of FMD tolerability, as defined by the occurrence of G3-G4 adverse events, or serious adverse events (SAEs)
Correlation between FMD-induced changes in serum metabolites and changes in PBMCs | 3 years
  Correlation between FMD-induced changes in serum metabolites and changes in PBMCs, their activation status, and characteristics of tumor cell and immune infiltrate.
Correlation between FMD-induced metabolic and immunological changes | 3 years
  Correlation between FMD-induced metabolic and immunological changes with patient diet evaluated at study enrollment through food diaries.

CONTACTS AND LOCATIONS:
Overall Officials: Filippo De Braud, Professor, Principal Investigator — Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Italy
Locations (1):
- Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hanahan D, Weinberg RA. Hallmarks of cancer: the next generation. Cell. 2011 Mar 4;144(5):646-74. doi: 10.1016/j.cell.2011.02.013. PMID 21376230
- [Background] Vernieri C, Casola S, Foiani M, Pietrantonio F, de Braud F, Longo V. Targeting Cancer Metabolism: Dietary and Pharmacologic Interventions. Cancer Discov. 2016 Dec;6(12):1315-1333. doi: 10.1158/2159-8290.CD-16-0615. Epub 2016 Nov 21. PMID 27872127
- [Background] Vander Heiden MG, Cantley LC, Thompson CB. Understanding the Warburg effect: the metabolic requirements of cell proliferation. Science. 2009 May 22;324(5930):1029-33. doi: 10.1126/science.1160809. PMID 19460998
- [Background] Locasale JW, Grassian AR, Melman T, Lyssiotis CA, Mattaini KR, Bass AJ, Heffron G, Metallo CM, Muranen T, Sharfi H, Sasaki AT, Anastasiou D, Mullarky E, Vokes NI, Sasaki M, Beroukhim R, Stephanopoulos G, Ligon AH, Meyerson M, Richardson AL, Chin L, Wagner G, Asara JM, Brugge JS, Cantley LC, Vander Heiden MG. Phosphoglycerate dehydrogenase diverts glycolytic flux and contributes to oncogenesis. Nat Genet. 2011 Jul 31;43(9):869-74. doi: 10.1038/ng.890. PMID 21804546
- [Background] Mankoff DA, Eary JF, Link JM, Muzi M, Rajendran JG, Spence AM, Krohn KA. Tumor-specific positron emission tomography imaging in patients: [18F] fluorodeoxyglucose and beyond. Clin Cancer Res. 2007 Jun 15;13(12):3460-9. doi: 10.1158/1078-0432.CCR-07-0074. PMID 17575208
- [Background] Sullivan LB, Gui DY, Hosios AM, Bush LN, Freinkman E, Vander Heiden MG. Supporting Aspartate Biosynthesis Is an Essential Function of Respiration in Proliferating Cells. Cell. 2015 Jul 30;162(3):552-63. doi: 10.1016/j.cell.2015.07.017. PMID 26232225
- [Background] Menendez JA, Lupu R. Fatty acid synthase and the lipogenic phenotype in cancer pathogenesis. Nat Rev Cancer. 2007 Oct;7(10):763-77. doi: 10.1038/nrc2222. PMID 17882277
- [Background] Menendez JA, Vellon L, Mehmi I, Oza BP, Ropero S, Colomer R, Lupu R. Inhibition of fatty acid synthase (FAS) suppresses HER2/neu (erbB-2) oncogene overexpression in cancer cells. Proc Natl Acad Sci U S A. 2004 Jul 20;101(29):10715-20. doi: 10.1073/pnas.0403390101. Epub 2004 Jul 2. PMID 15235125
- [Background] Yang YA, Han WF, Morin PJ, Chrest FJ, Pizer ES. Activation of fatty acid synthesis during neoplastic transformation: role of mitogen-activated protein kinase and phosphatidylinositol 3-kinase. Exp Cell Res. 2002 Sep 10;279(1):80-90. doi: 10.1006/excr.2002.5600. PMID 12213216
- [Background] Larkin J, Chiarion-Sileni V, Gonzalez R, Grob JJ, Cowey CL, Lao CD, Schadendorf D, Dummer R, Smylie M, Rutkowski P, Ferrucci PF, Hill A, Wagstaff J, Carlino MS, Haanen JB, Maio M, Marquez-Rodas I, McArthur GA, Ascierto PA, Long GV, Callahan MK, Postow MA, Grossmann K, Sznol M, Dreno B, Bastholt L, Yang A, Rollin LM, Horak C, Hodi FS, Wolchok JD. Combined Nivolumab and Ipilimumab or Monotherapy in Untreated Melanoma. N Engl J Med. 2015 Jul 2;373(1):23-34. doi: 10.1056/NEJMoa1504030. Epub 2015 May 31. PMID 26027431
- [Background] Eggermont AM, Chiarion-Sileni V, Grob JJ, Dummer R, Wolchok JD, Schmidt H, Hamid O, Robert C, Ascierto PA, Richards JM, Lebbe C, Ferraresi V, Smylie M, Weber JS, Maio M, Bastholt L, Mortier L, Thomas L, Tahir S, Hauschild A, Hassel JC, Hodi FS, Taitt C, de Pril V, de Schaetzen G, Suciu S, Testori A. Prolonged Survival in Stage III Melanoma with Ipilimumab Adjuvant Therapy. N Engl J Med. 2016 Nov 10;375(19):1845-1855. doi: 10.1056/NEJMoa1611299. Epub 2016 Oct 7. PMID 27717298
- [Background] Lee C, Raffaghello L, Brandhorst S, Safdie FM, Bianchi G, Martin-Montalvo A, Pistoia V, Wei M, Hwang S, Merlino A, Emionite L, de Cabo R, Longo VD. Fasting cycles retard growth of tumors and sensitize a range of cancer cell types to chemotherapy. Sci Transl Med. 2012 Mar 7;4(124):124ra27. doi: 10.1126/scitranslmed.3003293. Epub 2012 Feb 8. PMID 22323820
- [Background] Brandhorst S, Wei M, Hwang S, Morgan TE, Longo VD. Short-term calorie and protein restriction provide partial protection from chemotoxicity but do not delay glioma progression. Exp Gerontol. 2013 Oct;48(10):1120-8. doi: 10.1016/j.exger.2013.02.016. Epub 2013 Feb 21. PMID 23454633
- [Background] Lee C, Safdie FM, Raffaghello L, Wei M, Madia F, Parrella E, Hwang D, Cohen P, Bianchi G, Longo VD. Reduced levels of IGF-I mediate differential protection of normal and cancer cells in response to fasting and improve chemotherapeutic index. Cancer Res. 2010 Feb 15;70(4):1564-72. doi: 10.1158/0008-5472.CAN-09-3228. Epub 2010 Feb 9. PMID 20145127
- [Background] Safdie FM, Dorff T, Quinn D, Fontana L, Wei M, Lee C, Cohen P, Longo VD. Fasting and cancer treatment in humans: A case series report. Aging (Albany NY). 2009 Dec 31;1(12):988-1007. doi: 10.18632/aging.100114. PMID 20157582
- [Background] de Groot S, Vreeswijk MP, Welters MJ, Gravesteijn G, Boei JJ, Jochems A, Houtsma D, Putter H, van der Hoeven JJ, Nortier JW, Pijl H, Kroep JR. The effects of short-term fasting on tolerance to (neo) adjuvant chemotherapy in HER2-negative breast cancer patients: a randomized pilot study. BMC Cancer. 2015 Oct 5;15:652. doi: 10.1186/s12885-015-1663-5. PMID 26438237
- [Background] Dorff TB, Groshen S, Garcia A, Shah M, Tsao-Wei D, Pham H, Cheng CW, Brandhorst S, Cohen P, Wei M, Longo V, Quinn DI. Safety and feasibility of fasting in combination with platinum-based chemotherapy. BMC Cancer. 2016 Jun 10;16:360. doi: 10.1186/s12885-016-2370-6. PMID 27282289
- [Background] Cheng CW, Adams GB, Perin L, Wei M, Zhou X, Lam BS, Da Sacco S, Mirisola M, Quinn DI, Dorff TB, Kopchick JJ, Longo VD. Prolonged fasting reduces IGF-1/PKA to promote hematopoietic-stem-cell-based regeneration and reverse immunosuppression. Cell Stem Cell. 2014 Jun 5;14(6):810-23. doi: 10.1016/j.stem.2014.04.014. PMID 24905167
- [Background] Brandhorst S, Choi IY, Wei M, Cheng CW, Sedrakyan S, Navarrete G, Dubeau L, Yap LP, Park R, Vinciguerra M, Di Biase S, Mirzaei H, Mirisola MG, Childress P, Ji L, Groshen S, Penna F, Odetti P, Perin L, Conti PS, Ikeno Y, Kennedy BK, Cohen P, Morgan TE, Dorff TB, Longo VD. A Periodic Diet that Mimics Fasting Promotes Multi-System Regeneration, Enhanced Cognitive Performance, and Healthspan. Cell Metab. 2015 Jul 7;22(1):86-99. doi: 10.1016/j.cmet.2015.05.012. Epub 2015 Jun 18. PMID 26094889
- [Background] Di Biase S, Lee C, Brandhorst S, Manes B, Buono R, Cheng CW, Cacciottolo M, Martin-Montalvo A, de Cabo R, Wei M, Morgan TE, Longo VD. Fasting-Mimicking Diet Reduces HO-1 to Promote T Cell-Mediated Tumor Cytotoxicity. Cancer Cell. 2016 Jul 11;30(1):136-146. doi: 10.1016/j.ccell.2016.06.005. PMID 27411588

DOCUMENTS (1):
  • Study Protocol (2017-09-10): https://cdn.clinicaltrials.gov/large-docs/82/NCT03454282/Prot_000.pdf